CLINICAL TRIAL: NCT00166842
Title: Effects of Conversion From Sirolimus Oral Solution to Tablets in Renal Transplant Recipients.
Brief Title: Sirolimus Blood Concentrations on Conversion From Oral Solution to Tablets
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 910506; NTUH S92
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2005-09-14 (Estimated); Status verified 2002-07

CONDITIONS: Transplantation; Kidney Transplantation; Immunosuppression
Keywords: Pharmacokinetics; Sirolimus; Cyclosporine; Tacrolimus; Immunosuppressive Agents; Immunosuppression; Transplantation; Kidney Transplantation
MeSH Terms: interventions — Sirolimus; Cyclosporine; Tacrolimus

INTERVENTIONS:
Drug: sirolimus, cyclosporine, tacrolimus

SUMMARY:
The purpose of this study is to understand the pharmacokinetics of sirolimus tablets in different regimens in newly renal transplant patients, and the effect of dosage form conversion on the concentration of sirolimus in stable renal transplant patients. So that we can design a better tacrolimus or cyclosporine/sirolimus/steroid dose regimen for Taiwanese.

DETAILED DESCRIPTION:
Sirolimus tablets will be available more than one year after the launch of sirolimus solution. Most patients on sirolimus solution will use sirolimus tablet instead.

The purpose of this study is to understand the pharmacokinetics of sirolimus tablets in different regimens in newly renal transplant patients, and the effect of dosage form conversion on the concentration of sirolimus in stable renal transplant patients. So that we can design a better tacrolimus or cyclosporine/sirolimus/steroid dose regimen for Taiwanese.

ELIGIBILITY:
Inclusion Criteria:

* ages of 18 and 65, renal transplant patients

Exclusion Criteria:

* pregnancy, tuberculosis, hepatitis B or C carrier status, human immunodeficiency virus-positive status, retransplantation or multiorgan transplantation, or history of rheumatoid arthritis before transplantation

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2002-09

PRIMARY OUTCOMES:
Pharmacokinetics of sirolimus tablets in different regimens in de novo renal transplant patients
Effect of dosage form conversion on sirolimus concentration in stable renal transplant patients.

SECONDARY OUTCOMES:
Effectiveness of different sirolimus dose regimens in rejection prevention

CONTACTS AND LOCATIONS:
Overall Officials: Po-Huang Lee, MD PhD, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Result] Wu FL, Tsai MK, Sun SW, Chen RR, Huang JD, Lee PH. Effects of conversion from sirolimus oral solution to tablets in stable Taiwanese renal transplant recipients. J Formos Med Assoc. 2005 Jan;104(1):22-8. PMID 15660173